CLINICAL TRIAL: NCT04254679
Title: Opioid-free Analgesia After Outpatient General Surgery: A Pilot Randomized Controlled Trial
Brief Title: Pilot Trial: Postoperative Opioid-free Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Society of American Gastrointestinal and Endoscopic Surgeons (Other)
Responsible Party: Principal Investigator, Julio F Fiore Jr, Assitant Professor (McGill), McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUHC REB 2020-5965
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Outpatient Surgery; Abdominal Surgery; Breast Surgery
Keywords: Opioids; Surgery; Postoperative Period; Postoperative Pain; Analgesia; Pain Management
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Analgesics, Opioid; Analgesics, Non-Narcotic

STUDY DESIGN:
Intervention Model Description: This study will be a parallel, two-group, assessor-blind, pilot randomized trial.
Who Masked: Outcomes Assessor
Masking Description: Patient-reported outcomes and treatment adherence data will be collected via self-administered electronic questionnaires distributed using REDCap (http://project-redcap.org/) and completed by patients via smartphone, tablet or personal computer. Electronic outcome data will be transmitted directly to the REDCap database and verified by a blinded assessor. Adherence data will be verified by unblinded study staff. Patients who are not computer savvy, have limited access or prefer non-electronic assessment will complete the questionnaires via telephone interviews with a blinded assessor; in this case, data will be recorded in paper forms and subsequently transferred to the REDCap database. Outcome data that are not patient-reported (e.g. postoperative complications, unplanned healthcare utilization, chronic opioid use), will be obtained from medical records by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid analgesia (Experimental)
  Interventions: Drug: Opioid analgesics
- Opioid-free analgesia (Active Comparator)
  Interventions: Drug: Non-opioid analgesics

INTERVENTIONS:
Drug: Opioid analgesics — Current standard of care in the participating centers Prescription of around-the-clock non-opioid analgesics (acetaminophen and/or NSAIDs/COX-2) and a supply of opioids to be used as a rescue in case of breakthrough pain.
  The specific round-the-clock analgesia and rescue opioid regimens will be determined by the patient's primary surgeon considering the surgical procedure, comorbidities and patient's preference.
  Arms: Opioid analgesia
Drug: Non-opioid analgesics — Prescription of around-the-clock non-opioid analgesics (acetaminophen alone or combined with NSAIDs/COX-2).
  The specific non-opioid analgesia regimens will be determined by the patient's primary surgeon considering the surgical procedure, comorbidities and patient's preference.
  Arms: Opioid-free analgesia

SUMMARY:
North America is facing an opioid epidemic fueled by surgeons, who are the second largest subgroup of physicians involved in opioid prescribing. Surgery often serves as the initial event for opioid-naïve patients to obtain a prescription for opioids and spiral into misuse and addiction. From the perspective of perioperative care clinicians, the answer to the opioid crisis may be using opioid-free analgesia. However, the number of comparative studies in this field is limited and existing small trials do not reflect current standards of care in North America. Lack of evidence means that the decision to prescribe opioids after outpatient surgery largely depends on surgeon preference and healthcare culture. Hence, there is an urgent need for a robust randomized controlled trial (RCT) to guide clinical decision-making. The feasibility and optimal design of this RCT should be informed by a pilot trial. The overarching goal of this pilot RCT is to investigate the feasibility of conducting a full-scale RCT to assess the comparative-effectiveness of opioid versus opioid-free analgesia after outpatient general surgery.

DETAILED DESCRIPTION:
This study will be a pragmatic, parallel, two-group, assessor-blind, pilot RCT. The investigators aim to recruit 80 adult patients at two tertiary hospitals in Montreal. Eligibility criteria will span outpatient procedures in abdominal and breast surgery. Patients are randomized on a 1:1 ratio to treatment with either opioid (standard care) or without opioid (only non-opioid analgesics). Patients will be followed up for 3 months after surgery; postoperative day (POD) 1 to POD 7 and at 2, 3 and 4 weeks after surgery, and at 3 months. Assessments will include postoperative pain, physical and mental function, adverse drug events, prolonged opioid use and opioid misuse. Feasibility outcomes will include the number of patients screened, consented and randomized, adherence with treatment and completion of follow-up. Data from this pilot study will inform the calculation of sample size requirements for the full-scale RCT. An embedded qualitative study will be conducted to help optimize trial design based on clinicians' and patients' perspective.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>18 yo) undergoing outpatient surgery

* Abdominal surgery (i.e. cholecystectomies, hernia repairs, ovarian cystectomies, salpingectomies)
* Breast surgery (i.e. lumpectomies, partial and complete mastectomies, axillary node dissections)

Exclusion Criteria:

All patients

* Intraoperative or early postoperative complications (i.e. diagnosed in the Post-Anesthesia Care Unit (PACU)) that require postoperative hospital stay
* Contraindications to any of the drugs used in the trial
* Difficult to be reached after surgery
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Do U, El-Kefraoui C, Pook M, Balvardi S, Barone N, Nguyen-Powanda P, Lee L, Baldini G, Feldman LS, Fiore JF Jr; McGill Better Opioid Prescribing Collaboration; Alhashemi M, Antoun A, Barkun JS, Brecht KM, Chaudhury PK, Deckelbaum D, Di Lena E, Dumitra S, Elhaj H, Fata P, Fleiszer D, Fried GM, Grushka J, Kaneva P, Khwaja K, Lapointe-Gagner M, McKendy KM, Meguerditchian AN, Meterissian SH, Montgomery H, Rajabiyazdi F, Safa N, Touma N, Tremblay F. Feasibility of Prospectively Comparing Opioid Analgesia With Opioid-Free Analgesia After Outpatient General Surgery: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2221430. doi: 10.1001/jamanetworkopen.2022.21430. PMID 35849399

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Started | 42 | 39
Completed | 39 | 37
Not Completed | 3 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Excluded owing to intraoperative complication requiring hospital stay | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Analgesia | Opioid-free Analgesia | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (15.1) | 56.8 (14) | 55.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 15 | 11 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 39 | 37 | 76
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.4 (4.7) | 28.8 (8.7) | 27.6 (7)
BMI >= 30.0 [Count of Participants; unit: Participants] | 7 | 11 | 18
American Society of Anesthesiology score I [Count of Participants; unit: Participants] — Classified based on the ASA classification chart:
  ASA I Definition - A person in good health. (e.g., a person who doesn't smoke tobacco products and minimally uses alcohol.)
  Participants | 6 | 9 | 15
American Society of Anesthesiology score II [Count of Participants; unit: Participants] — Classified based on the ASA classification chart:
  ASA II Definition -A mild but well-managed or treated condition. (e.g., a person who is pregnant, has a mild lung condition, may smoke tobacco products or drinks alcohol socially or has overweight.)
  Participants | 25 | 28 | 53
American Society of Anesthesiology score III [Count of Participants; unit: Participants] — Classified based on the ASA classification chart:
  ASA III Definition - A serious condition that has an impact on a person's overall health. (e.g., A person who has a BMI greater than 40, alcohol use disorder or an implanted pacemaker.)
  Participants | 2 | 6 | 8
Risk of opioid abuse score (SD) [Mean (Standard Deviation); unit: units on a scale] — Potential for opioid misuse was assessed by the Screener and Opioid Assessment for Patients With Pain Short Form (5-item) questionnaire. The total score ranges from 0 to 20 and a score ≥ 4 indicates a likely high risk of opioid misuse after prescription.
  units on a scale | 2 (1.6) | 1.8 (1.7) | 1.9 (1.6)
Risk of opioid abuse score ≥4 [Count of Participants; unit: Participants] — Potential for opioid misuse was assessed by the Screener and Opioid Assessment for Patients With Pain Short Form (5-item) questionnaire. The total score ranges from 0 to 20 and a score ≥ 4 indicates a likely high risk of opioid misuse after prescription.
  Participants | 4 | 5 | 9
Pain catastrophizing score, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — This 13-item questionnaire (5-point scale, 0= "not at all", 4= "all the time") aims to quantify an individual's tendency to magnify the threat value of pain and to feel helpless in its presence.
  Scoring algorithms provide a total pain catastrophizing score (range 0-52, best-worst), as well as subscale scores (rumination, magnification and helplessness).
  units on a scale | 13.5 (10.7) | 13.6 (11) | 13.6 (10.7)
Employed, including self-employed [Count of Participants; unit: Participants] | 24 | 20 | 44
Retired [Count of Participants; unit: Participants] | 9 | 11 | 20
Homemaker [Count of Participants; unit: Participants] | 2 | 0 | 2
Student [Count of Participants; unit: Participants] | 0 | 1 | 1
Unemployed [Count of Participants; unit: Participants] | 1 | 4 | 5
Unable to work, receiving disability pension [Count of Participants; unit: Participants] | 3 | 1 | 4
Current smoker [Count of Participants; unit: Participants] | 8 | 5 | 13
Prerandomization treatment group preference: Unsure or no preference [Count of Participants; unit: Participants] | 13 | 15 | 28
Prerandomization treatment group preference: Opioid medication group [Count of Participants; unit: Participants] | 7 | 4 | 11
Prerandomization treatment group preference: Opioid-free medication group [Count of Participants; unit: Participants] | 19 | 18 | 37
Prerandomization perceptions of opioid-free analgesia: Very Effective [Count of Participants; unit: Participants] | 8 | 15 | 23
Prerandomization perceptions of opioid-free analgesia: Somewhat Effective [Count of Participants; unit: Participants] | 17 | 11 | 28
Prerandomization perceptions of opioid-free analgesia: Not effective [Count of Participants; unit: Participants] | 0 | 2 | 2
Prerandomization perceptions of opioid-free analgesia: No specific expectation [Count of Participants; unit: Participants] | 14 | 9 | 23
Abdominal Surgery [Count of Participants; unit: Participants] | 20 | 20 | 40
Laparoscopic appendectomy [Count of Participants; unit: Participants] | 0 | 1 | 1
Laparoscopic cholecystectomy [Count of Participants; unit: Participants] | 3 | 6 | 9
Laparoscopic inguinal hernia repair [Count of Participants; unit: Participants] | 8 | 1 | 9
Open inguinal hernia repair [Count of Participants; unit: Participants] | 8 | 9 | 17
Open umbilical hernia repair [Count of Participants; unit: Participants] | 1 | 2 | 3
Open incisional hernia repair [Count of Participants; unit: Participants] | 0 | 1 | 1
Breast surgery [Count of Participants; unit: Participants] | 19 | 17 | 36
Partial mastectomy [Count of Participants; unit: Participants] | 4 | 10 | 14
Partial mastectomy with sentinel node biopsy [Count of Participants; unit: Participants] | 7 | 4 | 11
Partial mastectomy with axillary node dissection [Count of Participants; unit: Participants] | 4 | 2 | 6
Partial mastectomy with sentinel node biopsy and reconstruction [Count of Participants; unit: Participants] | 0 | 1 | 1
Total mastectomy with sentinel node biopsy [Count of Participants; unit: Participants] | 2 | 0 | 2
Total mastectomy with sentinel node biopsy and reconstruction [Count of Participants; unit: Participants] | 1 | 0 | 1
Total mastectomy with axillary node dissection and reconstruction [Count of Participants; unit: Participants] | 1 | 0 | 1
Received intraoperative regional analgesia [Count of Participants; unit: Participants] | 31 | 26 | 57
Peripheral nerve block [Count of Participants; unit: Participants] | 5 | 6 | 11
Wound infiltration [Count of Participants; unit: Participants] | 31 | 26 | 57
Duration of surgery [Mean (Standard Deviation); unit: min] | 97 (39) | 84 (51) | 91 (45)
Amount of opioids received in the PACU [Mean (Standard Deviation); unit: MME] | 18 (14) | 25 (21) | 21 (18)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Screened Participants Who Were Eligible to Participate in the Study
Description: At least 70% of patients undergoing the outpatient general surgery procedures of interest (screened participants) are eligible to be randomized.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Total Number of Screened Patients: Total number of patients undergoing outpatient general surgery procedures.
Arm/Group | Total Number of Screened Patients
Number analyzed (Participants) | 224
Participants | 163

2. Primary Outcome: Percentage of Surgeons Agreeing and Adhering to Patient Randomization
Description: At least 90% of the surgeons who agreed to have their patients randomized comply with the agreement (i.e. not change their minds).
Time Frame: 4 months
Population: *Providers were not considered as enrolled participants but did contribute to this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Total Number of Surgeons: The total number of surgeons conducting general surgery procedures at the intended sites.
Arm/Group | Total Number of Surgeons
Number analyzed (Participants) | 15
Participants | 15

3. Primary Outcome: Percentage of Eligible Patients Agreeing to Participate
Description: At least 50% of eligible patients agree to participate in the study and are randomized.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Total Number of Screened Patients
Number analyzed (Participants) | 168
Participants | 93

4. Primary Outcome: Percentage of Randomized Patients Complying With Allocated Treatment
Description: At least 80% of the randomized patients comply with their allocated treatment (i.e. will take their pain medications as prescribed).
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Opioid Analgesia: The total number of patients included in the opioid analgesia arm
- Opioid-free Analgesia: The total number of patients included in the opioid-free analgesia arm
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
Participants | 39 | 36

5. Primary Outcome: Percentage of Randomized Patients Completing the 30-day Postoperative Outcome Assessment
Description: At least 80% of the randomized patients complete outcome assessment at 30 days after surgery.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
Participants | 39 | 34

6. Primary Outcome: Percentage of Missing Data Among All Questionnaires Distributed to Patients Who Completed the Assessments
Description: Among all questionnaires distributed to patients who complete outcome assessments, the proportion of missing data (i.e. non-response to questionnaires) is less than 10%.
Time Frame: 4 months
Population: As this is a feasibility trial, the feasibility outcomes were predetermined based on the protocol and were assessed and reported using the entire participant sample.
Measure: Count of Units; unit: Questionnaires
Units Other Than Participants: Questionnaires
Groups:
- Total Study Participants: Total number of patients who completed the outcome assessments.
Arm/Group | Total Study Participants
Number analyzed (Participants) | 76
Number analyzed (Questionnaires) | 3724
Questionnaires | 37

7. Primary Outcome: Percentage of Missing Data Among All Questionnaire Items Distributed to Patients Who Completed the Assessments
Description: Among patients who complete outcome assessments, the proportion of missing data is less than 10% (i.e. non-response to specific questionnaire items).
Time Frame: 4 months
Population: as for outcome 6
Measure: Count of Units; unit: Questionnaire Items
Units Other Than Participants: Questionnaire Items
Groups:
- Questionnaires: Total number of items in the questionnaire distributed to study participants in the study
Arm/Group | Questionnaires
Number analyzed (Participants) | 76
Number analyzed (Questionnaire Items) | 32256
Questionnaire Items | 33

8. Secondary Outcome: Postoperative Pain
Description: Measured using the Brief Pain Inventory Short-Form, which addresses pain severity and interference in the last 24 hours. Scores range from 0 to 10; higher scores represent worse pain outcomes.
Time Frame: 30 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
score on a scale
  Baseline Severity Scale score | 0.9 (1.7) | 1 (2)
  Post Operative Day (POD) 1 Severity Scale score | 2.8 (2.2) | 3 (1.7)
  POD2 Severity Scale score | 2.7 (2.3) | 2.6 (2.1)
  POD3 Severity Scale score | 2.1 (2) | 1.7 (1.8)
  POD4 Severity Scale score | 1.6 (1.7) | 1.4 (1.7)
  POD5 Severity Scale score | 1.3 (1.7) | 1.1 (1.3)
  POD6 Severity Scale score | 1.2 (1.5) | 1.1 (1.4)
  POD7 Severity Scale score | 1.1 (1.6) | 0.9 (1.2)
  Post Operative Week (POW) 2 Severity Scale score | 0.9 (1.4) | 0.4 (0.8)
  POW3 Severity Scale score | 0.5 (1) | 0.4 (0.8)
  POW4 Severity Scale score | 0.5 (1.3) | 0.3 (0.8)
  Baseline Interference Scale score | 0.9 (1.9) | 0.7 (1.7)
  POD 1 Interference Scale score | 3 (3.1) | 3.3 (2.1)
  POD 2 Interference Scale score | 2.4 (2.5) | 2.3 (2)
  POD 3 Interference Scale score | 1.9 (2.5) | 1.8 (1.9)
  POD 4 Interference Scale score | 1.6 (2.6) | 1.4 (1.9)
  POD 5 Interference Scale score | 1.1 (1.9) | 1 (1.7)
  POD 6 Interference Scale score | 1.2 (2) | 0.8 (1.5)
  POD 7 Interference Scale score | 1.1 (2) | 1 (1.9)
  POW 2 Interference Scale score | 1 (1.7) | 0.5 (1.5)
  POW 3 Interference Scale score | 0.6 (1.5) | 0.4 (1.2)
  POW 4 Interference Scale score | 0.2 (0.6) | 0.1 (0.6)

9. Secondary Outcome: Time to Stopping Pain Medication
Description: The time to the first report of stopping the use of pain medication.
Time Frame: 30 days.
Measure: Mean (Standard Deviation); unit: days postoperative
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
days postoperative | 9 (9) | 9 (7.9)

10. Secondary Outcome: Postoperative Health Status
Description: Measured using the PROMIS-29 questionnaire, which assesses 7 domains of health (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference). Norm-based scores are calculated for each domain, such that a score of 50 represents the mean of the general population (standard deviation=10). Higher scores represent more of the domain being measured.
Time Frame: Weeks 1, 2, 3 and 4 after surgery.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
T-score
  Physical functioning Baseline | 50.2 (8.3) | 50.8 (8.6)
  Physical functioning Post Operative Week (POW) 1 | 44.9 (8.3) | 44.1 (9.1)
  Physical functioning POW 2 | 47.2 (7.5) | 47.9 (8.1)
  Physical functioning POW 3 | 49.6 (7.7) | 50.6 (7.3)
  Physical functioning POW 4 | 52.1 (7) | 51.5 (7.2)
  Social participation Baseline | 55 (9.4) | 52.9 (8.7)
  Social participation POW 1 | 49.6 (9.6) | 47.3 (10.4)
  Social participation POW 2 | 54.5 (8.8) | 54.4 (8.3)
  Social participation POW 3 | 56.5 (8) | 55.6 (8.6)
  Social participation POW 4 | 57.2 (8.4) | 56.6 (8.4)
  Anxiety Baseline | 53.3 (9.9) | 53 (8.5)
  Anxiety POW 1 | 46.4 (8.4) | 48.6 (8)
  Anxiety POW 2 | 45.9 (8.1) | 44.7 (6.9)
  Anxiety POW 3 | 44.4 (6.4) | 43.2 (5.6)
  Anxiety POW 4 | 44.5 (6.7) | 44.4 (6.7)
  Depression Baseline | 47.1 (8.7) | 48 (8.2)
  Depression POW 1 | 45.6 (6.8) | 46.2 (7.2)
  Depression POW 2 | 45.1 (6.7) | 43.6 (5.8)
  Depression POW 3 | 44.7 (6.4) | 43.7 (5)
  Depression POW 4 | 44.1 (5.3) | 44.3 (6)
  Pain interference Baseline | 49.1 (9) | 48.4 (8.9)
  Pain interference POW 1 | 55.7 (8.3) | 55.5 (9.1)
  Pain interference POW 2 | 50.5 (8.9) | 49.9 (7.1)
  POW 3 | 48.5 (7.6) | 46.5 (7.3)
  POW 4 | 45.9 (6.8) | 46.7 (7.1)
  Sleep disturbance Baseline | 46.8 (9.8) | 49.3 (8.6)
  Sleep disturbance POW 1 | 47.1 (8.5) | 47.4 (9.1)
  Sleep disturbance POW 2 | 45.2 (7.5) | 46.9 (9)
  Sleep disturbance POW 3 | 45 (8.3) | 46.1 (9.3)
  Sleep disturbance POW 4 | 43.6 (8.5) | 44.3 (9.3)
  Fatigue Baseline | 45.9 (9.5) | 47.7 (10)
  Fatigue POW 1 | 48.4 (9.4) | 50.2 (11.2)
  Fatigue POW 2 | 43 (9.6) | 44.6 (10.3)
  Fatigue POW 3 | 41.8 (8.2) | 42.4 (9.9)
  Fatigue POW 4 | 40.9 (7.7) | 42.2 (9.8)

11. Secondary Outcome: Opioid Side-effects
Description: Measured using the Perioperative Opioid-Related Symptom Distress Scale, which records symptom distress due to common adverse effects experienced by patients who receive opioids to relieve postoperative pain.
  The reported rates indicate the number of reported events per period of evaluation.
Time Frame: Postoperative days 1 to 7, weeks 2, 3 and 4 after surgery
Measure: Number; unit: Number of reported events
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
Number of reported events
  Constipation : 7-day rate (any event) | 16 | 12
  Constipation : 7-day rate (clinically meaningful event) | 4 | 2
  Constipation : 30-day rate (any event) | 18 | 15
  Constipation : 30-day rate (clinically meaningful event) | 7 | 3
  Nausa : 7-day rate (any event) | 8 | 6
  Nausa : 7-day rate (clinically meaningful event) | 1 | 1
  Nausa : 30-day rate (any event) | 9 | 8
  Nausa : 30-day rate (clinically meaningful event) | 1 | 1
  Vomiting : 7-day rate (any event) | 3 | 1
  Vomiting : 7-day rate (clinically meaningful event) | 0 | 1
  Vomiting : 30-day rate (any event) | 6 | 1
  Vomiting : 30-day rate (clinically meaningful event) | 0 | 1
  Itching : 7-day rate (any event) | 13 | 7
  Itching : 7-day rate (clinically meaningful event) | 1 | 1
  Itching : 30-day rate (any event) | 15 | 15
  Itching : 30-day rate (clinically meaningful event) | 1 | 2
  Fatigue : 7-day rate (any event) | 31 | 28
  Fatigue : 7-day rate (clinically meaningful event) | 2 | 5
  Fatigue : 30-day rate (any event) | 32 | 30
  Fatigue : 30-day rate (clinically meaningful event) | 3 | 11
  Drowsiness : 7-day rate (any event) | 14 | 13
  Drowsiness : 7-day rate (clinically meaningful event) | 0 | 1
  Drowsiness : 30-day rate (any event) | 14 | 13
  Drowsiness : 30-day rate (clinically meaningful event) | 0 | 1
  Dizziness : 7-day rate (any event) | 7 | 6
  Dizziness : 7-day rate (clinically meaningful event) | 0 | 1
  Dizziness : 30-day rate (any event) | 8 | 7
  Dizziness : 30-day rate (clinically meaningful event) | 0 | 1
  Inability to concentrate : 7-day rate (any event) | 6 | 11
  Inability to concentrate : 7-day rate (clinically meaningful event) | 1 | 2
  Inability to concentrate : 30-day rate (any event) | 8 | 11
  Inability to concentrate : 30-day rate (clinically meaningful event) | 1 | 2
  Difficulty with urination : 7-day rate (any event) | 3 | 3
  Difficulty with urination : 7-day rate (clinically meaningful event) | 1 | 1
  Difficulty with urination : 30-day rate (any event) | 4 | 4
  Difficulty with urination : 30-day rate (clinically meaningful event) | 1 | 1
  Confusion : 7-day rate (any event) | 2 | 3
  Confusion : 7-day rate (clinically meaningful event) | 0 | 1
  Confusion : 30-day rate (any event) | 2 | 3
  Confusion : 30-day rate (clinically meaningful event) | 0 | 1

12. Secondary Outcome: Rate of Opioid Misuse
Description: Measured using the Prescription Opioid Misuse Index, which includes questions regarding excessive dose, frequency of use, need for early refills, feeling high from the medication, taking the medication due to stress and obtaining prescriptions from multiple physicians. Scores range from 0 to 6; an affirmative answer to >1 question indicates the patient exhibits prescription opioid misuse.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
score on a scale | 0.1 (0.4) | 0.1 (4)

13. Secondary Outcome: Postoperative Complications Classification
Description: Graded by severity using the Dindo-Clavien classification. This system grades complications according to the therapy needed for treatment (grades I to IV, best to worse).
  Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions.
  Grade II: Complications requiring drug treatments other than those allowed for Grade I complications; this includes blood transfusion and total parenteral nutrition (TPN) Grade III: Complications requiring surgical, endoscopic or radiological intervention Grade IIIa - intervention not under general anaesthetic Grade IIIb - intervention under general anaesthetic
Time Frame: 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
Participants
  I | 3 | 1
  II | 2 | 0
  IIIa/b | 1 | 1

14. Secondary Outcome: Rate of Unplanned Healthcare Utilization
Description: Emergency department visits, hospital readmissions.
Time Frame: 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
Participants
  Any | 6 | 1
  ED visit | 5 | 0
  Readmission | 1 | 1
  Outpatient clinic visit | 2 | 0

15. Secondary Outcome: Rate of Adverse Drug Events
Description: Obtained from spontaneous patient reporting (Trigger question "Did you have any significant medical problem related or unrelated to your surgery since the last study assessment?"). Events were coded using the MedDRA coding dictionary, graded by severity according to the Common Terminology Criteria for Adverse Events (CTCAE) and assessed for potential causality using the WHO/UMC system.
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
Participants
  Headache | 4 | 1
  Abdominal distention | 0 | 3
  Diarrhea | 1 | 2
  Postoperative wound infection | 2 | 0
  Cough | 1 | 1
  Urinary retention | 1 | 1
  Hypertention | 1 | 0
  Tachycardia | 1 | 0
  Breast haematoma | 1 | 0
  Productive cough | 0 | 1
  Dyspepsia | 0 | 1
  Ecchymosis | 1 | 0
  Hypoesthesia | 1 | 0
  Neuralgia | 1 | 0
  Oropharyngeal pain | 0 | 1
  Penile swelling | 0 | 1
  Testicular swelling | 0 | 1
  Seroma | 0 | 1
  Urinary tract infection | 0 | 1
  Cystitis | 0 | 1
  Peripheral neuropathy | 0 | 1

16. Secondary Outcome: Rate of Prolonged Opioid Use
Description: Filling of opioid prescriptions up to 3 months after surgery.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
Participants
  Post Operative Week (POW) 1 | 25 | 1
  POW 2 | 0 | 0
  POW 3 | 0 | 0
  POW 4 | 0 | 0
  POM 2 | 0 | 1
  POM 3 | 1 | 2

17. Secondary Outcome: Comprehensive Complication Index at 30-day
Description: Measured using the Comprehensive Complication Index score at 30 after surgery. The score ranges from 0 to 100; higher scores indicate greater severity of complications.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
Number analyzed (Participants) | 39 | 37
score on a scale | 2.6 (7.2) | 0.9 (4.5)

ADVERSE EVENTS:
Time Frame: The adverse events data were collected up to 30 days after surgery.
Description: Opioid side effects were identified by using the Perioperative Opioid-Related Symptom Distress Scale. Also, data regarding adverse drug events was obtained from spontaneous patient reporting and from data reported by clinicians in electronic medical records. Two independent clinicians coded adverse event data using the MedDRA coding dictionary. Disagreements regarding coding were resolved by consensus.
Arm/Group | Opioid Analgesia | Opioid-free Analgesia
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/39 | 1/37
Other Adverse Events (participants affected / at risk) | 14/39 | 16/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Analgesia (N=39) | Opioid-free Analgesia (N=37)
Breast Haematoma (Surgical and medical procedures) | 1 (1) | 0 (0)
Seroma (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Opioid Analgesia (N=39) | Opioid-free Analgesia (N=37)
Headache (General disorders) | 4 | 1
Abdominal distention (Surgical and medical procedures) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 2
Postoperative wound infection (Surgical and medical procedures) | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 3 — A clinically meaningful event as per the Perioperative Opioid-Related Symptom Distress Scale description.
Itching (General disorders) | 1 | 2 — A clinically meaningful event as per the Perioperative Opioid-Related Symptom Distress Scale description.
Fatigue (General disorders) | 3 | 11 — A clinically meaningful event as per the Perioperative Opioid-Related Symptom Distress Scale description.
Inability to concentrate (General disorders) | 1 | 2 — A clinically meaningful event as per the Perioperative Opioid-Related Symptom Distress Scale description.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT04254679/Prot_SAP_000.pdf